CLINICAL TRIAL: NCT00726479
Title: A Phase II, Randomised, Double-blind, Placebo-controlled and Parallel Group Study to Evaluate the Safety and Efficacy of Four Weeks Treatment of 7.5 mg b.i.d, 15 mg q.d and 15 mg b.i.d. BIBW 2948 BS (Inhalation Powder, Hard Capsule for HandiHaler®) in Patients With COPD Associated With Chronic Bronchitis.
Brief Title: Safety and Efficacy of 4-weeks Treatment of BIBW 2948 BS in Patients With Chronic Obstructive Bronchitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1219.4; EUDRACT2007-003742-15
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

INTERVENTIONS:
Drug: BIBW 2948 BS — 7.5 mg b.i.d, 15mg q.d, 15mg b.i.d

SUMMARY:
The primary objective of this study is to investigate the effect of 4-week treatment with 7.5 mg b.i.d, 15 mg q.d and 15 mg b.i.d. BIBW 2948 BS and placebo on cough and sputum as determined by the CASA-Q (Cough and Sputum Assessment Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. Male or female patients 40 years of age or older.
3. Patients must have a diagnosis of COPD defined by a post-bronchodilator FEV1 < 80% of predicted and FEV1 < 70% of FVC (to be obtained 30 minutes after administration of salbutamol HFA). Predicted normal values will be calculated according to ECSC (R94-1408).

   For Height measured in inches

   Males:

   FEV1 predicted (L) = 4.30 x (height (inches)/39.37) - 0.029 x age (yrs) - 2.49

   Females:

   FEV1 predicted (L) = 3.95 x [height (inches)/39.37] - 0.025 x age (yrs) - 2.60

   or Height measured in meters

   Males:

   FEV1 predicted (L) = 4.30 x [height (meters)] - 0.029 x age (yrs) - 2.49

   Females:

   FEV1 predicted (L) = 3.95 x [height (meters)] - 0.025 x age (yrs) - 2.60
4. Patients must have a diagnosis of chronic bronchitis symptoms i.e., cough and sputum expectoration on most days for at least three months in each of two consecutive years.
5. Patients must be a current or ex-smoker with a smoking history of sup or egal to 10 pack years (Patients who have never smoked cigarettes must be excluded).
6. Patients must be able to perform all specified procedures and able to maintain all necessary records during the study period as required in the protocol.
7. Patients must be able to inhale medication in a competent manner from the HandiHaler® device for BIBW 2948 BS.
8. Patients must be able to read and understand the questionnaires in the languages provided (English in the U.S., French in France and German in Germany).

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patients at risk because of participation in the study or may influence either the results of the study or the patient's ability to participate in the study.Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis if the abnormality defines a significant disease as defined in exclusion criteria No. 1.
2. Patients with an acute or chronic hepatitis or alpha one antitrypsin deficiency or other liver disease.
3. Patients with an aspartate aminotransferase (AST), alanine aminotransferase (ALT) 1.5 x the upper limit of the normal range will be excluded regardless of the clinical condition. A repeat laboratory evaluation will not be conducted in these patients.
4. Patients with history of asthma or allergic rhinitis.
5. Patients with history of post-nasal drip the last 3 months prior visit 1.
6. Patients with a clinical diagnosis of bronchiectasis.
7. Patients currently treated with expectorants and/or mucolytics drug.
8. Patients taking medications with known cough promoting side effects (e.g., angiotensin converting enzyme inhibitors or angiotensin II receptor blockers) that in the opinion of the investigator are causing symptoms of cough.
9. Patients with any respiratory tract infection or COPD exacerbation in the 30 days prior the visit 1 or during the 1-week period prior to visit 2 (visit 2 will not be postponed and the patient will be discontinued from the study).
10. Patients who have had any change in their respiratory medications within the last 6 weeks prior the visit 1.
11. Patients with a history of thoracotomy for other reasons should be evaluated as per Exclusion 1.
12. Patients with a history of gastroesophageal reflux disease that have changed medication (dose intensification or a change in therapy) to treat this disease within the 6 weeks prior the visit 1.
13. Patients with a history of cancer, other than treated basal cell carcinoma, within the last five years.
14. Women of childbearing potential or who have not been post-menopausal for a duration for at least 2 years and have not had a hysterectomy or tubal ligation procedure.
15. Participation in another trial with an investigational drug within 30 days or 6 half lives (whichever is greater) of the start of the study.
16. A known hypersensitivity to lactose or any other component of the inhalation capsule or any other components of the inhalation capsule delivery system.
17. Patients who are currently in a pulmonary rehabilitation program or who have completed a pulmonary rehabilitation program within four weeks prior the visit 1.
18. Patients with a significant history of significant alcohol or drug abuse.
19. Patients with previous participation in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be change in the Cough and Sputum PRO symptom domain scores from baseline (Visit 2) to the end of the 4 weeks treatment period. | 4 weeks

SECONDARY OUTCOMES:
Cough and Sputum PRO symptom domain scores Cough and Sputum PRO impact domain scores 24 hours sputum wet/dry weight and volume Cough frequency as recorded by electronic recording of thorax movement Interleukin 8 P. Level Cough and Sputum Rating Sc | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- United States (8):
  - 1219.4.01001 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1219.4.01007 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1219.4.01006 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1219.4.01002 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1219.4.01008 Boehringer Ingelheim Investigational Site, Rincon, Georgia
  - 1219.4.01003 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1219.4.01004 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1219.4.01005 Boehringer Ingelheim Investigational Site, Union, South Carolina
- France (10):
  - 1219.4.3306A Boehringer Ingelheim Investigational Site, Béthune
  - 1219.4.3306B Boehringer Ingelheim Investigational Site, Béthune
  - 1219.4.3302A Boehringer Ingelheim Investigational Site, Marseille
  - 1219.4.3303A Boehringer Ingelheim Investigational Site, Montpellier
  - 1219.4.3308A Boehringer Ingelheim Investigational Site, Nice
  - 1219.4.3307A Boehringer Ingelheim Investigational Site, Nîmes
  - 1219.4.3307B Boehringer Ingelheim Investigational Site, Nîmes
  - 1219.4.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1219.4.3305A Boehringer Ingelheim Investigational Site, Toulouse
  - 1219.4.3305B Boehringer Ingelheim Investigational Site, Toulouse
- Germany (6):
  - 1219.4.49003 Boehringer Ingelheim Investigational Site, Eisenach
  - 1219.4.49004 Boehringer Ingelheim Investigational Site, Hamburg
  - 1219.4.49001 Boehringer Ingelheim Investigational Site, Hanover
  - 1219.4.49006 Boehringer Ingelheim Investigational Site, Mainz
  - 1219.4.49005 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 1219.4.49002 Boehringer Ingelheim Investigational Site, Rüdersdorf